CLINICAL TRIAL: NCT04452071
Title: Gingival Crevicular Fluid Alkaline Phosphatase Activity as a Biomarker of Skeletal Maturation in Comparison to Modified Middle Phalanx of The Middle Finger (MP3) Method in a Sample of Growing Egyptian Females
Brief Title: Gingival Crevicular Fluid Alkaline Phosphatase as Skeletal Growth Indicator
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, sarah samir abdelrahman abelmaged, doctor, Cairo University
Other Study IDs: GCF ALP skeletal indicator
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Growth Indictaor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- prepubertal: patients born in 2012-2011
  Interventions: Radiation: periapical xray
- pubertal: patients born in 2010-2009-2008-2007
  Interventions: Radiation: periapical xray
- postpubertal: patients born in 2006-2005-2004-2003
  Interventions: Radiation: periapical xray

INTERVENTIONS:
Radiation: periapical xray — periapical xray on the middle phalanax of the middle finger

SUMMARY:
Determination of the pubertal growth spurt in Egyptian female patients using gingival crevicular fluid alkaline phosphatase

DETAILED DESCRIPTION:
assessment of the pubertal growth spurt in growing Egyptian female patients by using a simple, quick and easy method, through taking a gingival crevicular fluid alkaline phosphatase sample and measuring its concentration. Comparing the concentration of GCF ALP to the standardized middle phalanax of the middle finger MP3 we can predict if it can be an accurate and reliable method as skeletal growth indicator.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: only female subjects will be included.
2. Age between 7-16 years old
3. Intermediate or late mixed dentition and permanent dentition
4. Good general health with absence of any nutritional problems or bony disease
5. No usage of any anti-inflammatories or antibiotics in the month preceding the study
6. Fully erupted upper and lower central incisors for sample collection
7. Good gingival and periodontal health as indicated by Probing depth (PD) values that should not exceed 3 mm for the whole dentition.
8. Willingness to participate in the study and sign the informed consent form

Exclusion Criteria:

1. Male adolescent subjects
2. Periodontal and /or gingival disease
3. Systemic and/or bone disease

3. Growth abnormality

Ages: 7 Years to 16 Years | Sex: Female
Age Groups: Child
Gender Based: Yes — self representation of gender identity
Study Population: Egyptian female patients with age range from 7 to 16 years old
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
GCF ALP concentration | immediately after sample collection
  concentration of gingival crevicular fluid alkaline phosphatase
MP3 | immediately after taking x-rays
  periapical x-ray of the middle phalanax of the middle finger

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Manial, Egypt

REFERENCES:
- [Background] Perinetti G, Baccetti T, Contardo L, Di Lenarda R. Gingival crevicular fluid alkaline phosphatase activity as a non-invasive biomarker of skeletal maturation. Orthod Craniofac Res. 2011 Feb;14(1):44-50. doi: 10.1111/j.1601-6343.2010.01506.x. Epub 2010 Nov 23. PMID 21205168